CLINICAL TRIAL: NCT00351364
Title: The Effect of Leukotriene Receptor Blockade on Endothelial Function in Acute Coronary Syndrome Patients
Brief Title: Does Montelukast Have an Affect on the Function of the Artery in Patients With Heart Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Diffic;ulty recruiting
Sponsor: University of Calgary (Other)
Collaborators: Foothills Interventional Cardiology Group (Unknown)
Responsible Party: Principal Investigator, Todd Anderson, Director Libin Cardiovascular Institute, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18169
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: atherosclerosis; inflammation; leukotriene blockade; endothelial function
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Atherosclerosis; Inflammation | interventions — montelukast; Single Person

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Montelukast sodium (Active Comparator): Drug arm - Montelukast as a single dose 100 mg. To test the hypothesis of leukotriene inhibition.
  Interventions: Drug: Montelukast Sodium
- 2 (Placebo Comparator): No drug given - no placebo available. To compare with active drug.
  Interventions: Drug: Montelukast Sodium

INTERVENTIONS:
Drug: Montelukast Sodium — 100 mg P.O. One time only
  Other Names: singular

SUMMARY:
To evaluate the effect of the drug Montelukast on the brachial artery's function. By giving a drug like Montelukast, which blocks the effects of inflammation in the lungs arteries and controls asthma, we hope to see positive effects in other arteries such as in the heart.

DETAILED DESCRIPTION:
To measure the benefit of cysteinyl leukotriene blockade in favourably altering the pathophysiology of coronary artery disease. We hypothesize that patients admitted to hospital with acute coronary syndromes will have markedly abnormal endothelial function as measured by peripheral vasomotor responses to forearm ischemia. Patients with myocardial infarction and unstable angina have markedly increased renal excretion of the cysteinyl leukotriene metabolite LTE4 as observed in patients with asthma. Observations that coronary vessel tone is negatively affected by leukotrienes C4,D4 and E4 which influences the atherosclerotic process in these arteries. Studies that isolated the epicardial coronary arteries and challenged the vessels with an LTC4 and LTD4 concentration showed that coronary arterial myocytes were found to produce cysteinyl leukotrienes which lead to responsive vasoconstriction. The continued stimulus of vasoconstriction over time leads to endothelial dysfunction and disruption of the endothelium integrity which then leads to stressors that encourage a disease state and atherosclerosis.In this study we will specifically assess peripheral endothelial function by measuring brachial artery diameter changes and PAT responses to temporary forearm ischemia in patients that have had an acute coronary event before and after receiving Montelukast. As well we will measure leukotriene assays both in blood and urine .

ELIGIBILITY:
Inclusion Criteria:

* male or female age 18-80 years, diagnosis of acute coronary syndrome with one increased Troponin assay,chest pain or chest pain syndrome, stable on initial medical therapy, painfree x 6 hours prior to enrollment

Exclusion Criteria:

* STEMI, Q-wave MI, < 18years, women of childbearing potential, new LBBB, recurrent chest pain since hospitalization, IV nitroglycerine drip, hemodynamically unstable, history of asthma, history of liver disease or abnormal liver enzymes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The degree of brachial artery flow mediated dilation achieved compared between the control and interventional conditions. | 2 hours between baseline and follow up

SECONDARY OUTCOMES:
The degree of RH-PAT mediated dilation as a ratio of PVA during reactive hyperemia/ baseline PVA index will be compared between the control and Interventional conditions. | 2 hours between baseline and followup

CONTACTS AND LOCATIONS:
Overall Officials: David Goodhart, MD, Principal Investigator — Foothills Medical Center
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada